CLINICAL TRIAL: NCT07319039
Title: Breathlessness Patterns in Patients With Cancer, COPD and Heart Failure: an fMRI Feasibility Study
Acronym: BREACH-fMRI
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Lisa Hentsch, Doctor, University Hospital, Geneva
Other Study IDs: BREACH-fMRI
Record Dates: First submitted 2025-05-26; First posted 2026-01-06 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Heart Failure; Cancer; Volunteers
Keywords: Persistent dyspnea; Breathlessness; Palliative Medicine; Cerebral fMRI; Immersive virtual reality
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Heart Failure; Neoplasms; Dyspnea

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Patients and healthy volunteers who will have a cerebral fMRI
  Interventions: Other: Cerebral fMRI; Other: Immersive virtual reality

INTERVENTIONS:
Other: Cerebral fMRI — Neuroimaging data will be collected using a 3T Siemens Prisma MRI scanner (Prisma; Siemens, Erlangen, Germany) equipped with a 64-channel head coil. Functional T2*-weighted images will be acquired during the resting-state protocol. The sequences used will be gradient-echo planar imaging. Additionally, a single-band reference volume will be obtained prior to the functional acquisition, using the same parameters but without multiband (MB) acceleration, to assist in functional realignment and masking. A whole-brain T1-weighted multi-echo MPRAGE scan will also be performed with 1 mm isotropic resolution. three echo images were combined using the root-mean-square method.
Other: Immersive virtual reality — In collaboration with HypnoVR (HypnoVR, Strasbourg, France), patients will subsequently be provided with a visual immersion in a virtual world along with a scripted hypnotic voice track. HypnoVR's solution is certified as a medical device and has been studied in various medical contexts. The program will be adapted to run on its own dedicated PC instead of a (non-MRI compatible) HMD. As described in this protocol, the PL and the patients can select from a predefined set of virtual environments and choose the preferred voice-over script.

SUMMARY:
Dyspnea that persists despite optimal pathophysiological treatment is defined as persistent dyspnea.

Currently all brain functional magnetic resonance imaging (fMRI) studies conducted to evaluate breathlessness have done so using healthy volunteers or have concentrated on acute breathlessness. Little is known about chronic breathlessness patterns and their modulation by different triggers. Furthermore, it is currently assumed in the palliative care literature that patients suffering from different advanced and progressive diseases such as cancer, heart failure (HF) or chronic obstructive pulmonary disease (COPD) have the same triggers, perceptions and neurological pathways and thus require the same treatments/interventions (i.e. opioids as first line symptomatic pharmacologic treatment). However, it is now known that patients belonging to different disease groups do not necessarily benefit from opioids.

Aim of the study To assess the feasibility of identifying dyspnea patterns in different life-limiting conditions and to evaluate the effect of immersive virtual reality (IVR) on dyspnea using patient-reported-outcomes (PROMs).

Study procedure:

Patients with advanced chronic diseases such as cancer, COPD or HF suffering from dyspnea will undergo a brain fMRI in combination with an IVR intervention. The fMRI data will be reviewed to identify different patterns of dyspnea and the effect of IVR on dyspnea will be assessed through PROMs. Patients will be asked about the perceived burden of the study.

DETAILED DESCRIPTION:
Dyspnea that persists despite optimal pathophysiologic treatment is defined as persistent dyspnea.

Breathlessness, also defined as dyspnea, is a frequent symptom in patients with advanced and progressive diseases such as cancer, chronic obstructive pulmonary disease (COPD) and advanced heart failure (HF). In affected patients, breathlessness causes substantial suffering and is a major contributor to decreased quality of life.

Despite increasingly controversial data on the effectiveness of opioids in advanced disease, they are often prescribed according to expert opinion. It can be hypothesized that breathlessness is conveyed by a variety of different pathophysiologies resulting in various patterns of the central nervous system (CNS) signalling, requiring more than a one-size-fits-all answer to pharmacologic interventions (i.e. opioids).

In recent years, the healthcare industry has seen the development of immersive virtual reality therapies (IVR), also called "digital therapeutics". Immersive virtual reality is an interactive computer simulation that allows a person to be completely immersed within a three-dimensional virtual environment so that it has a real feeling of being in the virtual world. IVR has been used during magnetic resonance imaging (MRI), to reduce stress and anxiety perceived by patients who suffer from claustrophobia.

Functional MRI (fMRI) measures brain activity by detecting changes associated with blood flow. Studies conducted to evaluate breathlessness have done so using healthy volunteers, focusing on acute breathlessness or in the context of pulmonary rehabilitation. Little is known about persistent breathlessness patterns and their modulation by different triggers.

Aim of the study:

It is possible that breathlessness is experienced and centrally processed in different ways between different patients, related to: i) the underlying disease, ii) the triggers for breathlessness episodes, iii) differences in patient-reported multidimensional assessment items (i.e. perceived severity vs discomfort vs effort). This study aims to assess whether different patterns of breathlessness can be identified by fMRI technology.

Hypothesis:

The investigators hypothesize that it is possible for patients suffering from persistent breathlessness associated with COPD, heart failure and incurable and life-limiting cancer to undergo an fMRI and associated study interventions.

Primary objective:

To determine the feasibility and acceptability of an observational monocentric study using fMRI and IVR in breathlessness patients with COPD, heart failure and cancer.

Secondary objective:

To identify different breathlessness fMRI signals in different diseases (COPD, heart failure, cancer) and identify different types of breathlessness patterns using fMRI, IVR, and clinical parameters (including patient-reported-outcome measures (PROMs)).

Project design The investigators plan to conduct an observational study that involves the use of an fMRI and IVR. A feasibility study design was chosen because the included patients need particular consideration and the feasibility of the procedure (fMRI) needs to be evaluated.

Total number of participants: four patients with HF, four patients with COPD, four patients with cancer, four healthy volunteers.

Participants will be recruited at the outpatient palliative care clinic of the HUG (single center) on the basis of a screening of medical records of patients and the preverification of the inclusion and exclusion criteria mentioned above.

The healthy controls will be recruited from a convenience sampling of known healthy volunteers meeting the above criteria, from a similar age group, under no hierarchical influence from any member of the research team.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18 years and
* Followed by the outpatient palliative care clinic of the Geneva University Hospitals, Switzerland (HUG) and
* Breathlessness at rest > 2 and < 8 on the NRS (numeric rating scale 0 to 10) and
* Persistent breathlessness (persistent dyspnea for > 3 weeks despite adequate and maximal medication according to the pathology) and
* In a stable clinical condition, i.e., without an episode of acute cardiac, respiratory, and/or neurological failure leading to hospitalization in the previous 4 weeks and
* Diagnosis of either HF stage NYHA III-IV, or COPD with dyspnea on the modified MRC scale grade 3-4, or oncological disease with primary or secondary pulmonary involvement

Inclusion Criteria for Healthy Volunteers (Control Group)

* Age ≥ 18 years and
* No respiratory symptoms: dyspnea, cough, wheezing and
* No known pulmonary, cardiac, or oncological disease and
* Smoking status < 10 pack-years and
* No contraindication to fMRI (Appendix 3) and
* Ability to lie flat (supine position) and
* No diagnosed psychiatric illness (severe depression, severe anxiety, psychosis, other) or antipsychotic treatment deemed a contraindication for fMRI based on physician judgement and
* No neurological disorders according to neurological assessment, including diagnosed dementia (frontotemporal dementia, Alzheimer's disease, etc.), brain pathology (tumor, stroke, Parkinson's disease, etc.), or epilepsy and
* No claustrophobia, acrophobia, photophobia, severe hearing loss, and/or severe visual deficit and
* No contraindication to IVR (migraines, photosensitive epilepsy, vertigo)

Exclusion Criteria

* Breathlessness at rest ≥ 8 on the NRS (numeric rating scale 0 to 10)
* Contraindication to fMRI
* Inability to lie flat (supine position)
* Diagnosed psychiatric illness (severe depression, severe anxiety, psychosis, other) or antipsychotic treatment deemed a contraindication for fMRI based on physician judgement
* Neurological disorders according to neurological assessment, including diagnosed dementia (frontotemporal dementia, Alzheimer's disease, etc.), brain pathology (tumor, stroke, Parkinson's disease, etc.), or epilepsy
* Presence of claustrophobia, acrophobia, photophobia, severe hearing loss, and/or severe visual deficit
* Contraindication to IVR (migraines, photosensitive epilepsy, vertigo)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Followed by the outpatient palliative care clinic of the Geneva University Hospitals, Switzerland (HUG)
  Patient with a diagnosis of either HF stage NYHA III-IV or COPD with dyspnea on modified MRC scale grade 3-4 or oncological disease with either primary or secondary pulmonary location
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2025-08-26 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the study | 18 months after the beginning of the study
  Composite outcomes:
  1. Recruitment rate: proportion of eligible patients who consent to participate, calculated as the number of participants enrolled divided by the total number of eligible patients approached during the recruitment period. A recruitment rate ≥ 50% will be considered feasible.
  2. Retention rate: proportion of enrolled participants who complete the planned intervention (fMRI, vital signs, and study-associated questionnaires). A retention rate ≥ 70% will be considered acceptable.
  If both thresholds are met (recruitment rate and retention rate), progression to a larger observational study will be considered.

SECONDARY OUTCOMES:
Acceptability | 15 minutes after the procedure
  The acceptability for the patients is based on the intervention's perceived burden, evaluated on a 5-point Likert scale (1 meaning no burden, 5 the maximum possible burden), recorded within 15 minutes after the intervention, with a cutoff ≤ 3, indicating that the study was moderately burdensome.
Evolution of vital parameters | Before, during and 15 minutes after the fMRI
  Saturation in oxygen (SpO2) (%) (minimum and maximum values)
Evolution of vital parameters | Pre and 15 minutes after the fMRI
  Transcutaneous CO2 (ptCO2) (kPa) (minimum and maximum values)
Evolution of vital parameters | Pre and 15 minutes after the fMRI
  Respiratory rate over 1 minute (RR) (number/minute) (minimum and maximum values)
Evolution of dyspnea | Before, during and 15 minutes after the fMRI
  Evolution of the dyspnea form before the fMRI, during and 15 min after the procedure on a numerical scale from 0-10.
Evolution of vital parameters | Pre, during and 15 minutes after the fMRI
  Heart rate over 1 min (HR) (number/minute) (minimum and maximum values)
Claustrophobia questionnaire | 15 minutes after the procedure
  Claustrophobia questionnaire. This questionnaire has 26 questions scored from 0 (not at all anxious) to 4 (extremely anxious). It has been used to evaluate claustrophobia and its two components (fear of suffocation and fear of restriction) in patients undergoing MRI.

OTHER OUTCOMES:
fMRI parameters | During the procedure
  Percent signal change and latency of response in BOLD (blood-oxygen-level-dependent) signal change will be assessed in relevant brain regions, including the left precentral gyrus, left middle frontal gyrus, left insula, left amygdala, left hippocampus, medial orbitofrontal cortex, and brainstem regions.
fMRI parameters | During procedure
  Functional connectivity of the left and right anterior insula with multiple regions (anterior cingulate cortex)
fMRI parameters | During procedure
  Activation map of the brain areas with significant activity as derived from the BOLD signal
fMRI parameters | during procedure
  Peak amplitude (maximum change in BOLD signal during the trigger) will be assessed in relevant brain regions, including the left precentral gyrus, left middle frontal gyrus, left insula, left amygdala, left hippocampus, medial orbitofrontal cortex, and brainstem regions.
fMRI parameters | During procedure
  Cluster size of contiguous voxels with a significant activation
fMRI parameters | During procedure
  Measures of coupling between resting-state fMRI and respiration oscillations will be assessed in relevant brain regions, including the left precentral gyrus, left middle frontal gyrus, left insula, left amygdala, left hippocampus, medial orbitofrontal cortex, and brainstem regions, based on directed transfer analysis.
fMRI parameters | During procedure
  Perfusion MRI outcomes based on dynamic susceptibility contrast MR perfusion measurements: relative cerebral blood flow (rCBF) maps that allow determining rCBF in the left and right anterior insula

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Hentsch, Dr med, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University Hospitals, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tzourio-Mazoyer N, Landeau B, Papathanassiou D, Crivello F, Etard O, Delcroix N, Mazoyer B, Joliot M. Automated anatomical labeling of activations in SPM using a macroscopic anatomical parcellation of the MNI MRI single-subject brain. Neuroimage. 2002 Jan;15(1):273-89. doi: 10.1006/nimg.2001.0978. PMID 11771995
- [Background] Smallwood NE, Pascoe A, Wijsenbeek M, Russell AM, Holland AE, Romero L, Ekstrom M. Opioids for the palliation of symptoms in people with serious respiratory illness: a systematic review and meta-analysis. Eur Respir Rev. 2024 Oct 9;33(174):230265. doi: 10.1183/16000617.0265-2023. Print 2024 Oct. PMID 39384304
- [Background] Ekstrom M, Ferreira D, Chang S, Louw S, Johnson MJ, Eckert DJ, Fazekas B, Clark KJ, Agar MR, Currow DC; Australian National Palliative Care Clinical Studies Collaborative. Effect of Regular, Low-Dose, Extended-release Morphine on Chronic Breathlessness in Chronic Obstructive Pulmonary Disease: The BEAMS Randomized Clinical Trial. JAMA. 2022 Nov 22;328(20):2022-2032. doi: 10.1001/jama.2022.20206. PMID 36413230
- [Background] Finnegan SL, Browning M, Duff E, Harmer CJ, Reinecke A, Rahman NM, Pattinson KTS. Brain activity measured by functional brain imaging predicts breathlessness improvement during pulmonary rehabilitation. Thorax. 2023 Sep;78(9):852-859. doi: 10.1136/thorax-2022-218754. Epub 2022 Dec 26. PMID 36572534
- [Background] Yu L, De Mazancourt M, Hess A, Ashadi FR, Klein I, Mal H, Courbage M, Mangin L. Functional connectivity and information flow of the respiratory neural network in chronic obstructive pulmonary disease. Hum Brain Mapp. 2016 Aug;37(8):2736-54. doi: 10.1002/hbm.23205. Epub 2016 Apr 5. PMID 27059277
- [Background] Nakarada-Kordic I, Reay S, Bennett G, Kruse J, Lydon AM, Sim J. Can virtual reality simulation prepare patients for an MRI experience? Radiography (Lond). 2020 Aug;26(3):205-213. doi: 10.1016/j.radi.2019.11.004. Epub 2019 Nov 28. PMID 32052767
- [Background] Cataldo J, Collins S, Walker J, Shaw T. Use of virtual reality for MRI preparation and technologist education: A scoping review. J Med Imaging Radiat Sci. 2023 Mar;54(1):195-205. doi: 10.1016/j.jmir.2022.11.011. Epub 2022 Dec 30. PMID 36588009
- [Background] Garcia-Palacios A, Hoffman HG, Richards TR, Seibel EJ, Sharar SR. Use of virtual reality distraction to reduce claustrophobia symptoms during a mock magnetic resonance imaging brain scan: a case report. Cyberpsychol Behav. 2007 Jun;10(3):485-8. doi: 10.1089/cpb.2006.9926. PMID 17594277
- [Background] Kilic A, Brown A, Aras I, Hui R, Hare J, Hughes LD, McCracken LM. Using Virtual Technology for Fear of Medical Procedures: A Systematic Review of the Effectiveness of Virtual Reality-Based Interventions. Ann Behav Med. 2021 Oct 27;55(11):1062-1079. doi: 10.1093/abm/kaab016. PMID 33821879
- [Background] Wang S, Lim SH, Aloweni FBAB. Virtual reality interventions and the outcome measures of adult patients in acute care settings undergoing surgical procedures: An integrative review. J Adv Nurs. 2022 Mar;78(3):645-665. doi: 10.1111/jan.15065. Epub 2021 Oct 10. PMID 34633112
- [Background] O'Connor S, Mayne A, Hood B. Virtual Reality-Based Mindfulness for Chronic Pain Management: A Scoping Review. Pain Manag Nurs. 2022 Jun;23(3):359-369. doi: 10.1016/j.pmn.2022.03.013. Epub 2022 Apr 28. PMID 35491349
- [Background] Gaertner J, Fusi-Schmidhauser T, Stock S, Siemens W, Vennedey V. Effect of opioids for breathlessness in heart failure: a systematic review and meta-analysis. Heart. 2023 Jun 26;109(14):1064-1071. doi: 10.1136/heartjnl-2022-322074. PMID 36878671
- [Background] Morita T, Sakaguchi Y, Hirai K, Tsuneto S, Shima Y. Desire for death and requests to hasten death of Japanese terminally ill cancer patients receiving specialized inpatient palliative care. J Pain Symptom Manage. 2004 Jan;27(1):44-52. doi: 10.1016/j.jpainsymman.2003.05.001. PMID 14711468
- [Background] Morelot-Panzini C, Adler D, Aguilaniu B, Allard E, Bautin N, Beaumont M, Blanc FX, Chenivesse C, Dangers L, Delclaux C, Demoule A, Devillier P, Didier A, Georges M, Housset B, Janssens JP, Laveneziana P, Laviolette L, Muir JF, Ninot G, Perez T, Peiffer C, Schmidt M, Similowski T, Straus C, Taille C, Van Den Broecke S, Roche N; dyspnoea working group of the Societe de Pneumologie de Langue Francaise. Breathlessness despite optimal pathophysiological treatment: on the relevance of being chronic. Eur Respir J. 2017 Sep 27;50(3):1701159. doi: 10.1183/13993003.01159-2017. Print 2017 Sep. No abstract available. PMID 28954773
- [Background] Currow DC, Dal Grande E, Ferreira D, Johnson MJ, McCaffrey N, Ekstrom M. Chronic breathlessness associated with poorer physical and mental health-related quality of life (SF-12) across all adult age groups. Thorax. 2017 Dec;72(12):1151-1153. doi: 10.1136/thoraxjnl-2016-209908. Epub 2017 Mar 29. PMID 28356419
- [Background] Parshall MB, Schwartzstein RM, Adams L, Banzett RB, Manning HL, Bourbeau J, Calverley PM, Gift AG, Harver A, Lareau SC, Mahler DA, Meek PM, O'Donnell DE; American Thoracic Society Committee on Dyspnea. An official American Thoracic Society statement: update on the mechanisms, assessment, and management of dyspnea. Am J Respir Crit Care Med. 2012 Feb 15;185(4):435-52. doi: 10.1164/rccm.201111-2042ST. PMID 22336677